CLINICAL TRIAL: NCT05632276
Title: A Prospective, Multi Centre, Interventional, Non-comparator, Open Label Study to Demonstrate the Efficacy, Performance and Safety of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-Adhesive Dressings in the Management of Surgical and Traumatic Wounds
Acronym: MATILDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WC-22-440
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Surgical Wound; Trauma-related Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: A 4-week device intervention to demonstrate the efficacy, performance and safety of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-Adhesive dressings in the management of surgical and traumatic wounds
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ConvaFoam dressings (Other): Participants wounds will be assessed and will be allocated ConvaFoam Border, Silicone or Non-Adhesive dressing based upon the investigator's clinical judgment. participants will receive a dressing as part of a protocol of care for up to a period of 4 weeks
  Interventions: Device: ConvaFoam

INTERVENTIONS:
Device: ConvaFoam — ConvaFoam™ Border, ConvaFoam™ Non-Adhesive, and ConvaFoam™ Silicone dressings are designed to provide a moist wound healing environment. All participants will be assigned a dressing based upon clinical judgement for a maximum of 4 weeks with weekly assessments and dressing changes
  Other Names: ConvaFoam Silicone; ConvaFoam Border; ConvaFoam Non Adhesive

SUMMARY:
A prospective, multi centre, interventional, non-comparator, open label study to demonstrate the efficacy, performance and safety of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-Adhesive dressings in the management of surgical and traumatic wounds

DETAILED DESCRIPTION:
A prospective, multi centre, interventional, non-comparator, open label study to demonstrate the efficacy, performance and safety of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-Adhesive dressings in the management of surgical and traumatic wounds for up to 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients able and willing to provide informed consent
* Patients with Surgical wounds including incisional wounds including laparoscopic
* wounds and surgical wounds healing by secondary intention.
* Patients with Traumatic wounds
* Patients must be willing to attend visits as per schedule in protocol

Exclusion criteria:

* Patients with known allergies to any of the materials used in the dressing
* Patients who require any oxidising agents such as hydrogen peroxide or hypochlorite solutions.
* Patients, who in the opinion of the investigator, is considered unsuitable for any other reason
* Patients with wounds showing signs of infection on presentation or not resolving with the use of antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Demonstrate the efficacy of ConvaFoam ™ Border, ConvaFoam™ Non-Adhesive and ConvaFoam™ Silicone to manage the indicated acute wounds when used in accordance with the IFU | 4 weeks
  The efficacy will be measured by the dressings ability to manage exudate as demonstrated by:
  Lack of strikethrough
  Maintenance or improvement of peri-wound skin

SECONDARY OUTCOMES:
Demonstrate the performance of ConvaFoam™ Border, ConvaFoam™ Non-Adhesive and ConvaFoam™ Silicone to manage the indicated acute wounds when used in accordance with the IFU | 4 weeks
  Performance will be measured by:
  Wound healing as anticipated by primary or secondary intention
  Wear time
  Atraumatic removal
  Pain (pre application during application and on removal)
  Dressing comfort (patient satisfied with dressing comfort, able to resume activities of daily living)
  Ease of use
  Ease of removal
  Health Care Practitioner satisfaction
Demonstrate the safety of, ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-Adhesive dressings in the management of the indicated acute wounds when used in accordance with the IFU. | 4 weeks
  Safety will be measured by:
  Adverse reaction (including wound complications such as maceration, bleeding, blistering / protection of peri-wound edges / peri-wound skin integrity)
  Device Malfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Ozer, MD, Study Chair — Medical Director
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No